CLINICAL TRIAL: NCT01982721
Title: Evaluation of an Acceleration-Based Prosthetic Knee Locking Mechanism for Reducing the Risk of Falling in Transfemoral Amputees
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Collaborators: Dr. Sigal Portnoy (Unknown)
Responsible Party: Principal Investigator, Isabella Shvartz, Head of Rehabilitation Department, Hadassah Medical Organization
Other Study IDs: Roee_HMO-CTIL
Record Dates: First submitted 2013-10-30; First posted 2013-11-13 (Estimated); Last update posted 2016-03-31 (Estimated); Status verified 2016-03

CONDITIONS: Transfemoral Amputees

ARMS (2):
- Transfemoral amputees (Experimental): Locking mechanism for prosthetic knee (no trade mark provided)
  Interventions: Device: Locking mechanism for prosthetic knee
- Healthy volunteers (No Intervention)

INTERVENTIONS:
Device: Locking mechanism for prosthetic knee
  Arms: Transfemoral amputees

SUMMARY:
The investigators hypothesize that a new automatic prosthetic knee locking mechanism will improve gait characteristics during an induced controlled trip and reduce fear of falling.

ELIGIBILITY:
Inclusion Criteria:

* transfemoral amputees
* Independent ambulation with a prosthesis
* Full cognitive and cooperative ability to follow simple instructions
* No orthopaedic or neurologic impairments present, that are unrelated to the amputation at the time of the trial

Exclusion Criteria:

* Cognitive disorders preventing the subject from understanding the trial protocol, signing a consent form or following the researcher's instructions
* Orthopaedic or neurologic impairment, un-related to the amputation
* Pregnant woman
* Weight exceeding 100 kg

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2014-11; Primary Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
3D angles of the ankle, knee, hip and pelvis | One day

CONTACTS AND LOCATIONS:
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel